CLINICAL TRIAL: NCT06909838
Title: Radial Shockwave Therapy With ShockMaster 300® to Reduce Spasticity in Children With CP or Acquired Brain Injury: a Pilot Study
Brief Title: Radial Shockwave for Spasticity in Children With CP or ABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gymna Uniphy (Industry)
Collaborators: FRAME Jessa Ziekenhuis, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S68824
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Spasticity Due to Cerebral Palsy; Spasticity Post-Traumatic Brain Injury
Keywords: Extracorporeal shockwave therapy; shockwave therapy; shock wave therapy; children; radial shockwave therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (Active Comparator): Conventional physiotherapy plan
  Interventions: Other: Conventional treatment
- Shockwave and usual care (Experimental): All participants receive a 4-week rESWT intervention plan (4 sessions with a one week interval), as add-on to the conventional physiotherapy plan
  Interventions: Device: radial Extracorporeal shockwave therapy (rESWT); Other: Conventional treatment

INTERVENTIONS:
Device: radial Extracorporeal shockwave therapy (rESWT) — 4 rESWT interventions, with a one week interval, are added to the conventional treatment plan
  Arms: Shockwave and usual care
Other: Conventional treatment — Usual conventional therapy, including physiotherapy, ergotherapy, hippotherapy,..

SUMMARY:
The goal of this clinical trial is to determine if radial Extracorporeal shockwave therapy (rESWT) reduces spasticity in children with Cerbral Palsy (CP) or traumatic brain injury (TBI). The main questions it aims to answer are:

* Is it feasible to implement radial shockwave therapy in conventional physiotherapy plan in children with CP or TBI?
* Is it safe and effective to use rESWT for reducing spasticity in children with CP or TBI? Participants will receive a 4 week therapy intervention, as add on to the conventional physio (usual care), including one rESWT session per week for a total of 4 sessions.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy or acquired brain injury
* between 6-18 years old;
* gross motor function classification ≥2;
* experiencing spasticity in the lower limb (calf muscles, hip adductor muscles or hamstring muscles) and/or in the upper limb (biceps muscle, wrist flexor muscles, finger flexor muscles) with Modified Ashworth Scores (MAS) ≥1+.

Exclusion Criteria:

* recent (≤3 months) Botox injections or other recent (≤6 months) invasive intervention;
* local infections or wounds; neuropathy;
* severe organ dysfunction;
* severe psychosocial dysfunction that would not allow adhering to protocol;
* planned changes in medication dosage or medication scheme that might affect spasticity during a 4-month intervention and follow-up phase.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | Change from baseline to the end of intervention sessions at week 4
  The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion. The scale is validated for use in various clinical populations to measure spasticity. The MAS score varies form 0 (no increase in tone) up to 4 (limb rigid in flexion or extension).
Modified Ashworth Scale | Change from baseline to 3 months follow-up
  The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion. The scale is validated for use in various clinical populations to measure spasticity. The MAS score varies form 0 (no increase in tone) up to 4 (limb rigid in flexion or extension).

SECONDARY OUTCOMES:
Patient Specific Functional Scale | Change from baseline to the end of intervention sessions at week 4
  The PSFS focuses on the patient's opinion of their function, and requires the physiotherapist to ask the patient to list three activities that are limited by the condition for which they are seeking treatment. The current level of difficulty associated with the activities is rated on a 11 point scale, where "0" represents "unable to perform activity" and "10" represents "able to perform at prior level".
Patient Specific Functional Scale | Change from baseline to 3 months follow-up
  The PSFS focuses on the patient's opinion of their function, and requires the physiotherapist to ask the patient to list three activities that are limited by the condition for which they are seeking treatment. The current level of difficulty associated with the activities is rated on a 11 point scale, where "0" represents "unable to perform activity" and "10" represents "able to perform at prior level".
passive Range Of Motion | Change from baseline to the end of intervention sessions at week 4
  Passive range of motion (PROM) is the ROM that is achieved when a therapist exclusively causes movement of a joint and is usually the maximum range of motion that a joint can move. An increasing ROM in spasticity helps maintain or increase the extensibility of soft tissue and joints, reduces pain, improves function and can normalize muscle tone.
passive Range Of Motion | Change from baseline to 3 months follow-up
  Passive range of motion (PROM) is the ROM that is achieved when a therapist exclusively causes movement of a joint and is usually the maximum range of motion that a joint can move. An increasing ROM in spasticity helps maintain or increase the extensibility of soft tissue and joints, reduces pain, improves function and can normalize muscle tone.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aerssens, Pediatrician, Principal Investigator — MFC Sint Gerardus
Locations (1):
- Sint-Gerardus, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No